CLINICAL TRIAL: NCT01046383
Title: Effect of IMN1207 Versus Casein on, Weight Loss, Survival and Quality of Life in Non-small Cell Lung Cancer Patients During or Following Chemotherapy, Radiation or Surgery: A Multi-center Randomized, Double-blind Study - Phase III Trial
Brief Title: Effect of IMN1207 Versus Casein on Weight Loss, Survival and Quality of Life in Non-small Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slower than anticipated recruitment
Sponsor: Immunotec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMN1207-07
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2011-06

CONDITIONS: NON-SMALL CELL LUNG CANCER
Keywords: NON-SMALL CELL LUNG CANCER PATIENTS; WEIGHT LOSS; QUALITY OF LIFE; SURVIVAL; CHEMOTHERAPY; RADIOTHERAPY; SURGERY; CYSTEINE-RICH WHEY PROTEIN ISOLATE; IMN1207; CANCER-RELATED WASTING (CACHEXIA); BODY WEIGHT; NUTRITIONAL PROTEIN SUPPLEMENT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Weight Loss; Cachexia; Body Weight | interventions — Caseins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMN1207 (Experimental): Dietary Supplement: IMN1207
  Stratum A: CRP <40 mg/L and WBC < 11x109/L (i.e. subjects with relatively low levels of inflammation).
  Stratum B: CRP ≥ 40 mg/L and/or WBC ≥ 11x109/L (i.e. subjects with relatively high levels of inflammation.
  Interventions: Dietary Supplement: IMN1207
- Casein (Placebo Comparator): Dietary Supplement: Casein.
  Stratum A: CRP <40 mg/L and WBC < 11x109/L (i.e. subjects with relatively low levels of inflammation).
  Stratum B: CRP ≥ 40 mg/L and/or WBC ≥ 11x109/L (i.e. subjects with relatively high levels of inflammation.
  Interventions: Dietary Supplement: Casein

INTERVENTIONS:
Dietary Supplement: IMN1207 — 20 grams of IMN1207 per day for 40 weeks.
  Arms: IMN1207
Dietary Supplement: Casein — 20 grams of Casein per day for 40 weeks
  Arms: Casein

SUMMARY:
The primary aim of this IMN 1207 follow-up study is to confirm the effect of a cysteine-rich non-denatured whey protein isolate formulation IMN1207 (20g daily) versus casein (20 g daily) on the reversal of weight loss (cancer-related wasting) over a 40 week treatment period in non-small cell lung cancer patients with or without conventional therapy, i.e., chemotherapy or radiation. And to test the hypothesis that over a period of 66 weeks observation period which includes a 6 months follow-up period, increases the survival of these patients.

DETAILED DESCRIPTION:
This new IMN 1207 study is a follow-up study to the first IMN 1207 trial which was sponsored by Immunotec Inc during the last 3 years. The study revealed that the cysteine-rich whey protein isolate formulation IMN 1207 caused a significant reversal of weight loss (P <0.05) and a conspicuous increase in survival. The outcome of the first IMN 1207 study has been published in (Tozer RG, et al. Cysteine-Rich Protein Reverses Weight Loss in Lung Cancer Patients Receiving Chemotherapy or Radiotherapy. Antioxid Redox Signal. 2008 Feb; 10(2):395-402). PMID:18158761.

The purpose of this IMN 1207 follow-up study is to confirm the effect of a cysteine-rich non-denatured whey protein isolate formulation IMN1207 (20g daily) versus casein (20 g daily) on the reversal of weight loss (cancer-related wasting) over a 40 week treatment period in non-small cell lung cancer subjects with or without conventional therapy, i.e., chemotherapy or radiation. In addition, it is prospectively designed to test the hypothesis that, IMN1207 versus casein over a period of 66 weeks observation period which includes a 6 months follow-up period, increases the survival of these subjects. Also, the effect of IMN1207 on the quality of life in a defined subgroup of subjects will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer stage III or stage IV.
* Karnofsky performance status greater or equal to 70%.
* Expected participation in study for more than 3 months.
* Involuntary decrease in body weight of more than 3% over the 1-5 months period immediately preceding study entry.
* Age 18 or older.
* Serum creatine less or equal to 3.0mg/dL or 265 µmol/L.
* Total bilirubin in the normal range (0.2-1.2 mg/dL) SGPT equal to or less than 4 times the upper limit of normal.
* Reliable contraception (ovariectomy, hysterectomy, tubuligation for at least six months, oral contraceptive, barrier method, etc.) for women of child bearing potential.

Exclusion Criteria:

* History of angioedema or allergic reactions to any compound employed in this study.
* Pregnancy and lactating.
* Uncontrolled metastatic brain tumors.
* Milk protein intolerance.
* Subjects currently using N-acetylcysteine, alpha-lipoic acid supplements, or dry whey protein supplements.
* Presence of ascitis or edema according to principle investigator's clinical judgment.
* Significant anemia, as defined by the requirement of treatment with EPO.
* Subjects with either mild or soy allergy/intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the % change in body weight in the IMN1207 group compared to casein over a 40 weeks treatment period. | 40 weeks

SECONDARY OUTCOMES:
The survival/mortality over a 66 weeks observation period which includes a 6 months follow-up period | 66 weeks
The change in hand grip force. | 40 weeks
The change in Karnofsky performance status | 40 weeks
The assessment of the McGill QOL and the modified Edmonton Symptom Assessment Scale (ESAS). | 40 weeks
The 'repeated standing up/sitting down' test from the Simmonds Physical Performance assessment battery. | 40 weeks
The change in the plasma concentration of C-reactive protein (CRP). | 40 weeks
The change in lymphocyte counts. | 40 weeks
The change in the dose of chemotherapy (percent) or discontinuation of chemotherapy or interruption of radiation in response to patients' cachexia. | 40 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - CHUM - Hopital Notre Dame, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan